CLINICAL TRIAL: NCT04032002
Title: Involvement of Monocytic B1 and B2 Receptors in Inflammation and Chronic Vascular Disease in Patients With Hereditary Bradykinetic Angioedema
Acronym: MONOBRAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018/349/HP
Record Dates: First submitted 2019-07-22; First posted 2019-07-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hereditary Bradykinetic Angioedema
MeSH Terms: interventions — Space Flight; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients hereditary bradykinetic angioedema (Other)
  Interventions: Other: Explorations; Other: Blood samples
- healthy volunteers (Other)
  Interventions: Other: Explorations; Other: Blood samples

INTERVENTIONS:
Other: Explorations — On Day 1 vascular fonctions explorations performed
Other: Blood samples — On Day 1 35ml taken

SUMMARY:
The objective is to compare the gene expression of B1 and / or B2 monocyte receptors between patients with hereditary bradykinetic angioedema and control subjects.

ELIGIBILITY:
Inclusion Criteria (patients):

* Patient with inherited bradykinic angioedema due to quantitative or qualitative C1-inhibitor deficiencies, regardless of the frequency or severity of seizures and regardless of their background treatment, with the following diagnostic criteria:

  * C1-inhibitor rate <50% of normal
  * Repeated episodes characteristic of bradykinic angioedema
  * Hereditary nature of the disease.
* Person who read and understood the newsletter and signed the consent form
* Person affiliated with a social security scheme
* Effective contraception in women of childbearing age (negative pregnancy test). For postmenopausal women, a confirmatory diagnosis should be obtained (amenorrhea for at least 12 months before the inclusion visit).

Inclusion Criteria (volunteers):

* Person affiliated with a social security scheme
* Person who read and understood the newsletter and signed the consent form
* Effective contraception in women of childbearing age (negative pregnancy test). For postmenopausal women, a confirmation diagnosis should be obtained (amenorrhea for at least 12 months before the inclusion visit)

Exclusion Criteria (patients):

* Angioedema crisis less than 1 month old
* Chronic inflammatory disease such as rheumatoid arthritis or Crohn's disease.
* Acute infection in progress, with or without anti-infectious treatment
* Contraindication to the use of trinitrin:

  * Hypersensitivity to nitrates or to any of the excipients
  * shock, severe hypotension,
  * obstructive cardiomyopathy,
  * inferior court inferior myocardial infarction with right ventricular extension, except in case of evidence of left ventricular failure,
  * intracranial hypertension,
  * patient treated with sildenafil
* Pregnant or parturient or breastfeeding woman or lack of proven contraception
* Person deprived of liberty by an administrative or judicial decision or person placed under the protection of justice / sub-tutorship or curatorship
* Patient participating or having participated in another therapeutic trial within one week.

Exclusion Criteria (volunteers)

* Chronic inflammatory disease such as rheumatoid arthritis or Crohn's disease.
* Acute infection in progress, with or without anti-infectious treatment
* Contraindication to the use of trinitrin:

  * Hypersensitivity to nitrates or to any of the excipients
  * shock, severe hypotension,
  * obstructive cardiomyopathy,
  * inferior court inferior myocardial infarction with right ventricular extension, except in case of evidence of left ventricular failure,
  * intracranial hypertension,
  * patient treated with sildenafil
* Pregnant or parturient or breastfeeding woman or lack of proven contraception
* Person deprived of liberty by an administrative or judicial decision or person placed under the protection of justice / sub-tutorship or curatorship
* Person participating or having participated in another therapeutic trial within one week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
compare the gene expression of B1 and / or B2 monocyte receptors | Day 1
  compare between patients with hereditary bradykinetic angioedema and control subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- DRCI, Rouen, France

IPD SHARING:
Plan to Share IPD: No